CLINICAL TRIAL: NCT02405390
Title: Comparison of Head Motion in Pediatric Patients Endotracheally Intubated With Video Laryngoscopy (Storz C-Mac®) Versus Direct Laryngoscopy
Brief Title: Head Motion in Pediatric Patients Endotracheally Intubated With Video Laryngoscopy Versus Direct Laryngoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nicklaus Children's Hospital f/k/a Miami Children's Hospital (Other)
Collaborators: Florida International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20141780
Record Dates: First submitted 2015-02-17; First posted 2015-04-01 (Estimated); Results first posted 2017-06-12 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-03

CONDITIONS: Intubation; Difficult; Cervical Spine Injury
Keywords: Storz C-Mac®; Pediatric Airway; Cervical Spine Injury; Trauma Airway Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Video Laryngoscopy (Experimental): Some patients will be intubated with a video laryngoscope 'Storz C-Mac® laryngoscope'
  Interventions: Procedure: Video Laryngoscopy; Device: Storz C-Mac® laryngoscope
- Direct Laryngoscopy (Active Comparator): Some patients will be intubated with a direct (conventional) laryngoscope
  Interventions: Procedure: Direct Laryngoscopy; Device: Storz C-Mac® laryngoscope

INTERVENTIONS:
Procedure: Video Laryngoscopy — Head motion will be measured by using Polhemus Patriot™ electromagnetic tracking system
  Arms: Video Laryngoscopy
Procedure: Direct Laryngoscopy — Time for intubation will be measured from the laryngoscope entering the mouth to the endotracheal tube passing through the vocal cords
  Arms: Direct Laryngoscopy
Device: Storz C-Mac® laryngoscope

SUMMARY:
The purpose of this study is to evaluate if intubation with video laryngoscopy (VL) will result in less head motion and therefore less cervical motion when compared with direct laryngoscopy (DL).

The aim of the study is to determine the amount of head motion (extension, flexion and rotation) when using Storz C-Mac® video laryngoscopes and direct laryngoscopes. Secondarily, the study will also measure the number of attempts to properly intubate and the time required for intubation with either technique.

DETAILED DESCRIPTION:
Investigator initiated single site prospective and randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* patients being orally intubated in the Operating Room as per standard anesthesia procedures

Exclusion Criteria:

* previous history of cervical spine injury or surgery
* craniofacial abnormalities
* airway congenital abnormalities
* airway prior to surgery

Max Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2015-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Vargas Loayza, MD, Principal Investigator — Miami Children's Hospital Pediatric Emergency Medicine Fellow; Vincenzo Maniaci, MD, Study Director — Miami Children's Hospital Pediatric Emergency Medicine Attending
Locations (1):
- Miami Children's Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Miami Children's Hospital Research Institute Website — http://www.mch.com/for-medical-professionals/mch-research-institute.aspx

RESULTS

PARTICIPANT FLOW:
Groups:
- Video Laryngoscopy: Some patients will be intubated with a video laryngoscope
  Video Laryngoscopy: Head motion will be measured by using Polhemus Patriot™ electromagnetic tracking system
  Storz C-Mac® laryngoscope
- Direct Laryngoscopy: Some patients will be intubated with a direct (conventional) laryngoscope
  Direct Laryngoscopy: Time for intubation will be measured from the laryngoscope entering the mouth to the endotracheal tube passing through the vocal cords
  Storz C-Mac® laryngoscope
Period: Overall Study
Arm/Group | Video Laryngoscopy | Direct Laryngoscopy
Started | 46 | 46
Completed | 46 | 46
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Video Laryngoscopy | Direct Laryngoscopy | Total
Number analyzed (Participants) | 46 | 46 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.0 (1.8) | 4.07 (1.9) | 4.04 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 22 | 46
  Male | 22 | 24 | 46
Head Motion in degrees [Mean (Standard Deviation); unit: participants] — The primary measure was the degree of head motion which were maximum angles achieved with extension, flexion and rotation
  participants
    Extension | 17.7 (11.1) | 16.5 (9.5) | 17.05 (10.18)
    Flexion | 9.6 (8.0) | 8.3 (5.8) | 8.95 (6.9)
    Rotation Right | 9.1 (7.6) | 7.9 (6.6) | 8.48 (7.02)
    Rotation Left | 6.2 (4.4) | 6.5 (7.0) | 6.40 (5.76)

OUTCOME MEASURES:

1. Primary Outcome: Head Motion - Extension or Flexion
Description: Head motion will only be measured while the patient is being endotracheally intubated. Usually this takes less than one minute. No follow up after that.
Time Frame: During the process of intubation (less than one minute)
Measure: Mean (Standard Deviation); unit: degrees of extension
Groups:
- Video Laryngoscopy: Some patients will be intubated with a video laryngoscope. Head motion (extension, Flexion, Roation Right and Rotation Left) will be measured by using Polhemus Patriot™ electromagnetic tracking system
- Direct Laryngoscopy: Some patients will be intubated with a direct (conventional) laryngoscope. Head motion (extension, Flexion, Roation Right and Rotation Left) will be measured by using Polhemus Patriot™ electromagnetic tracking system
Arm/Group | Video Laryngoscopy | Direct Laryngoscopy
Number analyzed (Participants) | 45 | 46
degrees of extension | 16.5 (9.5) | 17.7 (11.1)

2. Secondary Outcome: Time for Intubation
Description: Time from when the laryngoscope blade enters the mouth until the endotracheal tube enters the vocal cords. No follow up after that.
Time Frame: During the process of intubation (less than one minute)
Measure: Mean (Standard Deviation); unit: second
Arm/Group | Video Laryngoscopy | Direct Laryngoscopy
Number analyzed (Participants) | 45 | 46
second | 25.8 (18.4) | 18.9 (10.8)

ADVERSE EVENTS:
Time Frame: Adverse events were considered from time of initiating intubation until successful tracheal intubation
Arm/Group | Video Laryngoscopy | Direct Laryngoscopy
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/46
Other Adverse Events (participants affected / at risk) | 0/46 | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes